CLINICAL TRIAL: NCT07343557
Title: Diagnostic Performance of Ultrasonographic Airway Measurements for Predicting Difficult Intubation in Adult Female Patients: A Prospective Observational Study
Brief Title: Ultrasound-Based Airway Assessment for Predicting Difficult Intubation in Adult Female Patients
Acronym: USG-AIRWAY
Status: Completed | Type: Observational
Sponsor: Adana City Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Uğur serkan Çitilcioğlu, Anesthesiologist, Adana City Training and Research Hospital
Other Study IDs: ADN-USG-AIRWAY-2025
Record Dates: First submitted 2025-12-29; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Difficult Intubation; Airway Assessment
Keywords: Airway Ultrasound; Tongue Thickness; Difficult Airway

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Airway Ultrasound Assessment Cohort: Adult female patients undergoing elective surgery in whom preoperative airway ultrasonography was performed for observational assessment of airway anatomy. No intervention was assigned as part of the study.

SUMMARY:
This prospective observational study aims to evaluate the ability of selected ultrasonographic airway measurements to predict difficult intubation in adult female patients undergoing elective surgery. Pre-induction airway ultrasonography will be performed to measure tongue thickness and anterior neck soft tissue-related parameters. These measurements will be compared with laryngoscopic findings during direct laryngoscopy. The results of this study may help identify practical and reliable ultrasound-based markers for preoperative airway assessment and improve patient safety.

DETAILED DESCRIPTION:
This is a prospective, single-center observational study conducted in adult female patients scheduled for elective surgery under general anesthesia. The study was performed at the University of Health Sciences Adana City Training and Research Hospital after approval by the institutional ethics committee.

Before induction of anesthesia, standardized ultrasonographic airway assessments were performed by an experienced anesthesiologist. Measurements included tongue thickness, the distance from the skin to the anterior commissure of the vocal cords, the distance from the skin to the hyoid bone, and the distance from the skin to the epiglottis. All measurements were obtained under static pre-induction conditions using portable ultrasound equipment.

Following anesthesia induction, direct laryngoscopy was performed, and laryngoscopic view was graded according to the Cormack-Lehane classification. Difficult intubation was defined based on predefined laryngoscopic criteria. Ultrasonographic measurements were then analyzed for their diagnostic performance in predicting difficult intubation.

The primary objective of the study was to determine the most informative ultrasonographic parameter for predicting difficult intubation in this population. Secondary objectives included comparing the relative diagnostic value of different ultrasound measurements and evaluating their potential role in routine preoperative airway assessment.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 18-65 years
* American Society of Anesthesiologists (ASA) physical status I-III physical status I-III
* Scheduled for elective surgery under general anesthesia requiring tracheal intubation
* Ability to provide informed consent

Exclusion Criteria:

* Body mass index ≥30 kg/m²
* Known history of difficult intubation
* Anatomical airway abnormalities or head and neck pathology
* Pregnancy
* Emergency surgery

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult female patients aged 18-65 years undergoing elective surgery under general anesthesia at a tertiary care hospital. Participants were non-pregnant and scheduled for non-emergency procedures.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2025-05-15 (Actual); Primary Completion 2025-12-15 (Actual); Study Completion 2025-12-15 (Actual)

PRIMARY OUTCOMES:
Incidence of Difficult Intubation | Perioperative
  Difficult intubation defined as Cormack-Lehane grade III or IV and/or the need for additional airway devices or techniques during tracheal intubation.

SECONDARY OUTCOMES:
Ultrasonographic Measurement of Tongue Thickness | Preoperative assessment
  Preoperative ultrasonographic measurement of tongue thickness performed in the suprahyoid region.
Ultrasonographic Measurement of Skin-to-Hyoid Bone Distance | Preoperative assessment
  Preoperative ultrasonographic measurement of the distance between the skin and the hyoid bone.
Ultrasonographic Measurement of Skin-to-Epiglottis Distance | Preoperative assessment
  Preoperative ultrasonographic measurement of the distance between the skin and the epiglottis.
Ultrasonographic Measurement of Distance from Skin to Anterior Commissure of the Vocal Cords | Preoperative assessment
  Preoperative ultrasonographic measurement of the distance from the skin to the anterior commissure of the vocal cords.

CONTACTS AND LOCATIONS:
Locations (1):
- Adana City Training and Research Hospital, Adana, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No